CLINICAL TRIAL: NCT04551248
Title: Post-marketing Safety Evaluation of 10 or 13-valent Pneumococcal Conjugate Vaccine in Children and 23-valent Pneumococcal Polysaccharide Vaccine in Elderly Adults.
Brief Title: Post-marketing Safety Evaluation of Pneumococcal Vaccines Among Children and Elderly Adults.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sungkyunkwan University (Other)
Collaborators: Government-wide R&D Fund project for infectious disease research (Unknown)
Responsible Party: Principal Investigator, Ju-Young Shin, Associate Professor, Sungkyunkwan University
Other Study IDs: SKKU-2020-PneV
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Pneumococcal Vaccine Adverse Reaction
Keywords: Pneumococcal conjugate vaccine; Pneumococcal polysaccharide vaccine; Adverse events following immunisation
MeSH Terms: interventions — 13-valent pneumococcal vaccine; PHiD-CV vaccine; 23-valent pneumococcal capsular polysaccharide vaccine; Influenza Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- PCV13 recipients (children): Children < 5 years who had received PCV10 or PCV13 from May, 2014 to December, 2018 under the national childhood immunization program in South Korea.
  Interventions: Biological: 10 or 13-valent pneumococcal conjugate vaccine
- PPSV23 recipients (elderly adults): Persons 65 years or older who had received at least one dose of PPSV23 between January, 2014 and December, 2018 under the national immunization program in South Korea.
  Interventions: Biological: 23-valent pneumococcal polysaccharide vaccine
- Influenza vaccine recipients (elderly adults): Persons 65 years or older who had received at least one dose of influenza vaccine (as comparator) between January, 2014 and December, 2018 under the national immunization program in South Korea.
  Interventions: Biological: Influenza vaccine

INTERVENTIONS:
Biological: 10 or 13-valent pneumococcal conjugate vaccine — a four-dose series that is indicated for use at 2, 4, 6, and 12 to 15 months of age.
  Other Names: Prevnar 13; Synflorix
  Groups: PCV13 recipients (children)
Biological: 23-valent pneumococcal polysaccharide vaccine — Single 0.5-mL dose administered intramuscularly or subcutaneously only.
  Other Names: Prodiax-23
  Groups: PPSV23 recipients (elderly adults)
Biological: Influenza vaccine — One dose of trivalent influenza vaccine in flu seasons.
  Groups: Influenza vaccine recipients (elderly adults)

SUMMARY:
The purpose of this observational study is to examine the risk of adverse events following vaccination with 10 or 13-valent pneumococcal conjugate vaccine (PCV10 or PCV13) among infants or children age <59 months and 23-valent pneumococcal polysaccharide vaccine (PPSV23) among adults age 65 years and older.

DETAILED DESCRIPTION:
The purpose of this observational study is to examine 1) the risk of adverse events (AEs) following vaccination with 10 or 13-valent pneumococcal conjugate vaccine (PCV10 or PCV13) among infants or children age <59 months using a self-controlled risk interval design and 2) the risk of AEs following vaccination with 23-valent pneumococcal polysaccharide vaccine (PPSV23) among adults age 65 years and older compared with influenza vaccine recipients using a cohort design. We will use the national health insurance database from the National Health Insurance Service (NHIS) linked with the national immunization program registry data from the Korea Centers for Diseases Control & Prevention (KCDC).

ELIGIBILITY:
Inclusion Criteria:

* Children < 5 years who had received PCV10 or PCV13 from May, 2014 to December, 2018.
* Persons 65 years or older who had received at least one dose of PPSV23 or influenza vaccine (as a comparator) between January, 2014 and December, 2018.

Exclusion Criteria:

* Persons who experienced outcomes of interest within 1 year before the date of vaccination.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Persons (children aged under 59 months and elderly adults aged 65 years and older) who received pneumococcal vaccines under the national immunization program.
Sampling Method: Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Relative risk of adverse events | 2014-2018
  1. the ratio of probability of adverse events occuring in the risk periods after vaccination with PCV10 or PCV13 versus the control periods in the self-controlled risk interval study design.
  2. the ratio of probability of adverse events occuring in the PPSV23 group versus the influenza vaccine (a comparator) group in the cohort study design.

CONTACTS AND LOCATIONS:
Overall Officials: Ju-Young Shin, PhD, Principal Investigator — Sungkyunkwan University
Locations (1):
- Sungkyunkwan University, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tseng HF, Sy LS, Qian L, Liu IA, Mercado C, Lewin B, Tartof SY, Nelson J, Jackson LA, Daley MF, Weintraub E, Klein NP, Belongia E, Liles EG, Jacobsen SJ. Pneumococcal Conjugate Vaccine Safety in Elderly Adults. Open Forum Infect Dis. 2018 May 2;5(6):ofy100. doi: 10.1093/ofid/ofy100. eCollection 2018 Jun. PMID 29977960
- [Background] Tseng HF, Sy LS, Liu IL, Qian L, Marcy SM, Weintraub E, Yih K, Baxter R, Glanz JM, Donahue J, Naleway A, Nordin J, Jacobsen SJ. Postlicensure surveillance for pre-specified adverse events following the 13-valent pneumococcal conjugate vaccine in children. Vaccine. 2013 May 24;31(22):2578-83. doi: 10.1016/j.vaccine.2013.03.040. Epub 2013 Apr 8. PMID 23579258
- [Background] Baker MA, Baer B, Kulldorff M, Zichittella L, Reindel R, DeLuccia S, Lipowicz H, Freitas K, Jin R, Yih WK. Kawasaki disease and 13-valent pneumococcal conjugate vaccination among young children: A self-controlled risk interval and cohort study with null results. PLoS Med. 2019 Jul 2;16(7):e1002844. doi: 10.1371/journal.pmed.1002844. eCollection 2019 Jul. PMID 31265459
- [Background] Miller ER, Moro PL, Cano M, Lewis P, Bryant-Genevier M, Shimabukuro TT. Post-licensure safety surveillance of 23-valent pneumococcal polysaccharide vaccine in the Vaccine Adverse Event Reporting System (VAERS), 1990-2013. Vaccine. 2016 May 27;34(25):2841-6. doi: 10.1016/j.vaccine.2016.04.021. Epub 2016 Apr 15. PMID 27087150
- [Background] Haber P, Arana J, Pilishvili T, Lewis P, Moro PL, Cano M. Post-licensure surveillance of 13-valent pneumococcal conjugate vaccine (PCV13) in adults aged ⩾19years old in the United States, Vaccine Adverse Event Reporting System (VAERS), June 1, 2012-December 31, 2015. Vaccine. 2016 Dec 7;34(50):6330-6334. doi: 10.1016/j.vaccine.2016.10.052. Epub 2016 Nov 9. PMID 27836437
- [Background] Trinh L, Macartney K, McIntyre P, Chiu C, Dey A, Menzies R. Investigating adverse events following immunisation with pneumococcal polysaccharide vaccine using electronic General Practice data. Vaccine. 2017 Mar 13;35(11):1524-1529. doi: 10.1016/j.vaccine.2017.01.063. Epub 2017 Feb 13. PMID 28202210